CLINICAL TRIAL: NCT06643949
Title: Takotsubo Italian Network: Italian Multicenter Observational Registry on Takostubo Syndrome
Brief Title: Italian Multicenter Observational Registry on Takostubo Syndrome
Acronym: TIN
Status: Active, not recruiting | Type: Observational
Sponsor: University of Molise (Other)
Responsible Party: Principal Investigator, Rodolfo Citro, Associate Professor, University of Molise
Other Study IDs: 141024
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Takotsubo Syndrome
Keywords: takotsubo; cardiomyopathy; cardiogenic shock; LVOTO; mitral regurgitation; heart failure
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Cardiomyopathies; Shock, Cardiogenic; Mitral Valve Insufficiency; Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — The registry will focus on the diagnostic and prognostic value of of echocardiographic features of patients with takotsubo syndrome

SUMMARY:
Takotsubo syndrome (TTS) has recently been described as an acquired form of cardiomyopathy whose pathophysiology is not yet well understood and mainly affects postmenopausal women. TTS or "broken heart" syndrome was first described in Japan in 1991. The Japanese term "tako-tsubo" means "polyp vessel" and describes the morphology of the left ventricular apex during systole in patients with this condition. The onset usually follows physical or emotional stress and mimics that of acute coronary syndrome (ACS) with a parade of symptoms, including chest pain, dyspnea, syncope, and nausea. Objective examination is often normal or otherwise nonspecific. ECG may document ST-T changes while echocardiogram shows areas of altered ventricular kinetics. Serum cardiac biomarkers may be increased. Currently, the gold standard method for the diagnosis of TTS is coronarography, which documents epicardial coronary arteries that are normal or free of critical lesions.

It is estimated that more than 2.5% of patients with a suspected diagnosis of ACS have TTS, and this number is probably underestimated. Although the prognosis of TTS is generally considered favorable, during the acute phase these patients can develop potentially fatal complications such as ventricular arrhythmias, cardiogenic shock, and heart rupture. Moreover, emerging scientific evidence sheds light on the need to adopt a dedicated diagnostic-therapeutic pathway for this type of patients.

The exact pathophysiology of TTS is still unknown and no large population studies or registries are currently available. Therefore, the purpose of the study is to better characterize the profile of this disease through the creation of a large registry.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with TTS in accordance with the InterTAK Diagnostic Criteria.

Exclusion Criteria:

* Age less than 18 years
* Myocarditis
* Acute coronary syndrome
* Myocardial infarction with non obstructive coronary arteries (MINOCA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with takotsubo syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 1 year
  Composite of acute heart failure, takotsubo recurrence and mortality.

IPD SHARING:
Plan to Share IPD: No